CLINICAL TRIAL: NCT06395233
Title: A Randomised Trial of the Effectiveness of Lottery, Assured and Combined Incentives on App Tracked Walking Behaviour Over 12 Weeks.
Brief Title: A Test of Different Incentives and How Effectively They Motivate Walking Behaviour
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-IHIREC
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Physical Inactivity
Keywords: Incentives; Physical activity; Apps; Digital Health; Health behaviour
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Three group randomised trial with no control
Who Masked: Participant, Investigator
Masking Description: Participants will be randomly allocated to their group and will not be aware of the incentives received by the other groups. Randomisation will be done by team setting up the study in the BetterPoints system and the principle investigator will only receive anonymised data and be blind to who has been allocated to each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group one: Assured Incentives (Experimental): Group 1: Assured (Points only): Participants will be able to earn 10 points for each 10 minutes of walking. Every minute will count, the participant does not have to walk for 10 consecutive minutes to receive the points. Once a person has accumulated 10 minutes of walking exercise, their points will be awarded. This will be capped at 40 points per day, i.e. the participant can earn 10 BetterPoints up to four times a day by doing 40 minutes of walking.
  Interventions: Device: BetterPoints App
- Group 2: Non Assured Incentives (Experimental): Group 2: Non-Assured (Lottery tickets only): Participants will be able to earn one lottery ticket for each 10 minutes of walking. This is accrued and awarded in the same way as the points condition. It is capped at four tickets per day.
  Interventions: Device: BetterPoints App
- Group 3: Combined (Experimental): Group 3: Combined (Combined points/tickets): Participants in group 3 will be able to earn 5 points and one lottery ticket for 10 minutes of walking. The daily lottery in this condition will be for 500 BetterPoints (rather than 1000 BetterPoints in group 2) and therefore each ticket will have an expected value (EV) of 5 BetterPoints. Participants will be able to earn points and tickets in this way for up to 40 minutes of walking per day.
  Interventions: Device: BetterPoints App

INTERVENTIONS:
Device: BetterPoints App — The BetterPoints app is a smartphone application that uses incentives and gamification to motivate physical activity.

SUMMARY:
This study aims to test the effectiveness of different types of incentives to motivate walking among people who use a tracker app. App users will be randomly allocated to three groups, Group 1 will received assured incentives in the form of points per minute of walking, Group 2 will received non-assured incentives in the form of prize draw tickets, one ticket per minute of walking and Group 3 will receive a combination of the two.

App-users will be invited to join the study and those who consent to joining will track their walking activity for 12 weeks using the BetterPoints app. Participants will also be asked to complete a survey at the start and end of the study period to assess motivation and responsiveness to reward.

At the end of the 12 weeks intervention period, changes in minutes of walking from the start of the study to three follow up time points will be assessed and compared between groups. Total minutes of walking will also be compared between groups. Differences in reported levels of autonomous motivation will be assessed between the start and end of the study and between groups.

DETAILED DESCRIPTION:
It is well established that physical activity reduces risks of common noncommunicable diseases. It is predicted that 65 million people in the United Kingdom will use a smartphone by 2025. With such reach, mobile apps show promise as an intervention to promote physical activity. Although systematic reviews suggest that financial incentives are effective in encouraging physical activity, their cost effectiveness at population level is still unknown. Studies combining apps and incentives suggest that the size of the incentive is not as important as the type, timing and content, which has implications for the affordability of interventions.

Two types of incentive used in apps are assured rewards that are earned per step/minute of physical activity, and lottery incentives, where activity is rewarded with more entries to prize draws. Whether assured or won in a lottery, rewards are in the form of a digital currency that can then be redeemed for shopping vouchers or donated to charity.

The cost of giving out assured rewards is dependent upon the number of users and their level of activity. With lottery-based approaches, costs can be fixed. That is, the prize(s) in the lottery are fixed regardless of the number of users and their activity. However, this means the expected win per user per activity falls with more users and users being more active. The evidence comparing lottery-based incentives is limited. Patel and colleagues compared different lottery conditions over 13 weeks and found that a combined approach offering an 18% chance of winning $5 and 1% chance of winning $50, was more effective than a high frequency-low pay out or jackpot. No research could be found that directly compared lottery-based approaches with assured incentives. This is the gap which the current trial aims to fill.

The present study aims to assess the efficacy of an assured vs lottery vs combined incentive in fostering physical activity. Insights from the study could help develop scalable, cost-effective interventions to improve public health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Existing users of the BetterPoints app. Not in sponsored programmes.

Exclusion Criteria:

BetterPoints app users who are under 18. BetterPoints app users who are enrolled in programmes sponsored by local authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-29 (Estimated); Primary Completion 2024-07-29 (Estimated); Study Completion 2024-07-29 (Estimated)

PRIMARY OUTCOMES:
Change in weekly minutes of walking from baseline | 12-weeks
  Baseline minutes of walking behaviour will be compared to follow up time points for the three groups. Minutes of walking will be measured using a GPS app. Baseline will be the two weeks of walking before the start of the intervention period. Follow up dates will be at four, eight and twelve weeks after the start of the intervention period.
Differences between groups in number of weekly minutes of walking achieved | 12-weeks
  Weekly minutes of walking will be plotted and visually inspected for differences between groups. Statistical differences in mean and median levels of walking at four, eight and twelve weeks will be tested. Proportional differences between groups in those reaching 150 minutes per week will be explored.

SECONDARY OUTCOMES:
Perceived motivation | 12-weeks
  Survey scores for autonomous motivation at the start and the end of the intervention period will be compared for changes within groups and differences in change between groups. The The shortened, 9-item version of the General Multifaceted Automaticity Scale (Boiché, J., et al, 2016. Shortened by Marchant et al, 2021) will be used. This is a Likert scale where participants are asked to indicate on a scale of one (I do not agree at all) to five (I totally agree) how much they agree with nine statements. Scoring: Sum and divide by 9. Low scores = low automaticity. High scores = high automaticity.
Reward responsiveness (RR) | 12-weeks
  RR will be measured at the start and end of the intervention period using the behavioural activation items from Gray's Behavioural Inhibition/Behaviour Activation scales(BIS/BAS) (Van den Berg et al, 2011. Carver C.S. 1994). Participants are asked to indicate the degree to which they agree (1) or disagree (4)with five statements using a Likert scale. RR will be assessed for changes over time by scoring the four items from the BAS in reverse i.e. a low score means highly reward responsive and a high score means low reward responsivness. Levels of RR will be explored as a predictors of levels of minutes of walking within and between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah McCarthy, MA, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available. Aggregated and anonymised data will be available upon reasonable request.